CLINICAL TRIAL: NCT03133728
Title: To Improve Rates of Antiretroviral Therapy Initiation for HIV-1 Infected Infants Through Point-of-Care Diagnosis
Brief Title: Diagnosis of HIV and Early Antiretroviral Therapy Initiation Among HIV-1 Infected Infants
Acronym: CDC Detect
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Albert Manasyan, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: UAB Neo 016
Record Dates: First submitted 2017-04-04; First posted 2017-04-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections; Hiv
Keywords: EID HIV; Early Infant Diagnosis; Point of Care; Infant; HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Intervention Group: The Investigators will visit each of the selected 3 clusters (i.e. 6 primary health clinics) to construct a retrospective cohort of high-risk HIV-infected women who entered the national PMTCT program and received the SOC between June 1, 2017 and May 31, 2018. Using existing data through the electronic health record information (SmartCare and LIMS), the investigators will gather individual-level retrospective data on high-risk Mother-Infant Pairs (MIPs) from PMTCT enrolment through the child's ART enrolment, initiation, and retention rate at 3 months.
- Post-Intervention Group: Study Research Assistants (RA) will review routine patient files and registers, augmented by existing electronic health record information, to identify a new cohort of high-risk Mother-Infant Pairs (MIPs) at each study site between the dates of June 1, 2019 and May 31, 2020. The outreach team will include, at a minimum, the study RA, a study peer, and an HIV counselor from the health facility, who will carry the Alere™ q HIV-1/2 Detect with them. When the outreach team contacts a high-risk MIP at community level, the team will approach the MIP for study screening, consent, and enrolment procedures. Study staff will ask the parent/guardian if the parent/guardian would like the IYC to be tested at their home, at a community health post, or other private space in the community. The IYC will be tested using both the Alere™ q HIV-1/2 Detect platform and a reflex DBS PCR test to evaluate performance of the POC platform in a mobile setting against the gold standard.
  Interventions: Diagnostic Test: Alere Q Testing

INTERVENTIONS:
Diagnostic Test: Alere Q Testing — Infants of intervention clinics will have heelprick-obtained blood tested by standard of care method (SOC) and Alere™ q HIV-1/2 Detect Test Point of Care testing onsite (i.e. community, household, or facility level). Point-of-care (POC) testing results will be available in 52 minutes. HIV-infected infants, based on the Alere Q test result, will start ART as soon as possible and start routine SOC visits at weeks 2, 4, 8, 12, 16, 20, 24, 36, and 48 post ART-initiation. Study data will be obtained on first 4 routine visits after ART initiation (3 months). Infants will return for results of DBS-based DNA PCR testing. Positive SOC infants remain on ART/study follow-up. Negative POC test/negative SOC infants will attend only routine care visits and continue on HIV prophylaxis per national guidelines. Discordant results require DNA PCR test, with positive results continuing ART, negative results being repeated for confirmation before discontinuation.
  Other Names: Alere™ q HIV-1/2 Detect Test Point-of-Care Testing
  Groups: Post-Intervention Group

SUMMARY:
The purpose of the study is to test the effect of the Alere™ q HIV-1/2 Detect (diagnostic assay) on uptake of HIV testing among HIV-exposed infants and young children, and health outcomes for HIV-infected infants and young children using a novel POC EID Community Model in Zambia. The study will also assess the feasibility of field implementation of this novel diagnostic tool and its acceptability among HIV-infected mothers and frontline health workers.

DETAILED DESCRIPTION:
The purpose of the study is to test the effect of the Alere™ q HIV-1/2 Detect (diagnostic assay) on uptake of HIV testing among HIV-exposed infants and young children, and health outcomes for HIV-infected infants and young children through a novel POC EID Community Model in Zambia. The study will also assess the feasibility of field implementation of this novel diagnostic tool and its acceptability among HIV-infected mothers and frontline health workers. The knowledge generated from this study will enable the Zambia Ministry of Health (MOH) to make informed policy decisions about the implementation and scale up of point of care (POC) diagnostic tools for early infant diagnosis and pediatric HIV treatment programs in Zambia and the region.

ELIGIBILITY:
Inclusion criteria include IYCs:

1. 0 days (at birth) - 17 months of age;
2. Probable or known HIV exposure documented through maternal sero-positivity or reactive infant HIV antibody test;
3. The IYC must be born to mothers who:

   1. attended ≥1 ANC visits without HIV testing; or
   2. delivered at home and did not return for post-natal care at a health facility, and thus the mother or their child were not tested for HIV; or
   3. were documented as HIV-infected but never initiated ART; or
   4. disengaged from HIV care after ART initiation/have not returned for ARV refills; or
   5. have not returned to the facility with their infant for initial EID testing or follow-up EID testing (after a negative test at birth or 6 weeks); or
   6. IYC not tested 6 weeks after cessation of breastfeeding.
4. With a parent/guardian ≥18 years of age, and willing and able to provide written informed consent in a study language (English, Nyanja, or Bemba).

Exclusion criteria include IYCs:

1. With documented age-appropriate, guideline-adherent receipt of DBS-based EID HIV PCR testing;
2. Already known to be HIV-infected / receiving ART.

Ages: 1 Minute to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-exposed infants and young children (up to 17 months of age)
Sampling Method: Non-Probability Sample
Enrollment: 1682 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Uptake of Antiretroviral Therapy (ART) among HIV-infected Infants and Young Children (IYC) | Baseline to 18 months
  Number of IYCs who were initiated on ARVs following a positive HIV test divided by the number of IYCs who tested positive for HIV.

SECONDARY OUTCOMES:
Age at first early infant HIV testing among HIV-exposed IYCs | Baseline to 18 months
  Average chronological ages of all IYCs when presenting for initial EID HIV testing.
3-month survival for HIV-infected IYC receiving ART | Baseline to 18 months
  Number of HIV-infected IYCs receiving ART who presented alive at 3 month visit divided by the total number of HIV-infected IYCs enrolled into ART.
3-month retention in care for HIV-infected IYC receiving ART | Baseline to 18 months
  Number of HIV-infected IYCs receiving ART who were retained in care at 6 month visit divided by the total number of HIV-infected IYCs enrolled in ART.
Time to ART initiation among HIV-infected IYCs using Alere™ q HIV-1/2 Detect | Baseline to 18 months
  Average time of ART initiation by IYCs who present for at initial HIV test following positive screening test within 17 months of age.
Describe knowledge of HIV-infected mothers regarding the Alere™ q HIV-1/2 Detect platform and POC EID Community Model | Baseline to 18 months
  A pre-defined set of questions will be asked to all the parent/guardians to evaluate their knowledge regarding the Alere ™ q HIV-1/2 Detect platform and POC EID Community Model. The Investigators will enroll a total of 20 parents/guardians of HIV-exposed IYC (3-4 will be recruited from each clinic) to participate in in-depth interviews (IDIs).
Describe attitudes of HIV-infected mothers regarding the Alere™ q HIV-1/2 Detect platform and POC EID Community Model | Baseline to 18 months
  A pre-defined set of questions will be asked to all the parent/guardians to evaluate their attitudes regarding the Alere ™ q HIV-1/2 Detect platform and POC EID Community Model. The Investigators will enroll a total of 20 parents/guardians of HIV-exposed IYC (3-4 will be recruited from each clinic) to participate in IDIs.
Describe preferences of HIV-infected mothers regarding the Alere™ q HIV-1/2 Detect platform and POC EID Community Model | Baseline to 18 months
  A pre-defined set of questions will be asked to all the parent/guardians to evaluate their knowledge regarding the Alere ™ q HIV-1/2 Detect platform and POC EID Community Model. The Investigators will enroll a total of 20 parents/guardians of HIV-exposed IYC (3-4 will be recruited from each clinic) to participate in IDIs.
Characterize feasibility of using the Alere™ q HIV-1/2 Detect platform and POC EID Community Model by the health care workers | Baseline to 18 months
  A pre-defined set of questions will be asked to all the healthcare providers to characterize the feasibility of using the Alere ™ q HIV-1/2 Detect platform and POC EID Community Model. The Investigators will enroll a total of 20 healthcare providers who have used the platform to participate in IDIs.
Characterize the acceptability of using the Alere™ q HIV-1/2 Detect platform and POC EID Community Model by the health care workers | Baseline to 18 months
  A pre-defined set of questions will be asked to all the healthcare providers to characterize the acceptability of using the Alere ™ q HIV-1/2 Detect platform and POC EID Community Model. The Investigators will enroll a total of 20 healthcare providers who have used the platform to participate in IDIs.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Manasyan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (6):
- Zambia (6):
  - George Primary Health Clinic, Lusaka
  - Kalingalinga Primary Health Clinic, Lusaka
  - Kamwala Primary Health Clinic, Lusaka
  - Makeni Primary Health Clinic, Lusaka
  - Matero Ref Primary Health Clinic, Lusaka
  - N'gombe Primary Health Clinic, Lusaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manasyan A, Tembo T, Dale H, Pry JM, Itoh M, Williamson D, Kapesa H, Derado J, Beard RS, Iyer S, Gass S, Mwila A, Herce ME. Differentiated community-based point-of-care early infant diagnosis to improve HIV diagnosis and ART initiation among infants and young children in Zambia: a quasi-experimental cohort study. BMJ Glob Health. 2025 Feb 20;10(2):e015759. doi: 10.1136/bmjgh-2024-015759. PMID 39979018